CLINICAL TRIAL: NCT07262073
Title: Prospective Randomized Controlled Study Comparing Peak Expiratory Flow (PEF) Changes After Robot-Assisted and Open Radical Prostatectomy
Brief Title: Comparison of Peak Expiratory Flow Changes After Robot-Assisted Versus Open Radical Prostatectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Betül Güven, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TABED1-25-1680
Record Dates: First submitted 2025-11-23; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer (CRPC); Peak Expiratory Flow
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open Radical Prostatectomy (Control Group) (Active Comparator): Patients undergoing open radical prostatectomy under standardized general anesthesia. No pneumoperitoneum or steep Trendelenburg position is applied.
  Interventions: Diagnostic Test: Surgical procedure: Robot-assisted laparoscopic radical prostatectomy
- Robot-Assisted Laparoscopic Radical Prostatectomy (Study Group) (Experimental): Patients undergoing robot-assisted laparoscopic radical prostatectomy (RALRP) under standardized general anesthesia, with carbon dioxide pneumoperitoneum and Trendelenburg positioning.
  Interventions: Diagnostic Test: Surgical procedure: Robot-assisted laparoscopic radical prostatectomy

INTERVENTIONS:
Diagnostic Test: Surgical procedure: Robot-assisted laparoscopic radical prostatectomy — RALRP will be performed with pneumoperitoneum (12-15 mmHg CO₂ insufflation) and 25-30° Trendelenburg position. Peak Expiratory Flow (PEF) will be measured preoperatively, 2 hours postoperatively, and 24 hours postoperatively using the same handheld peak flow meter.

SUMMARY:
This prospective, randomized controlled trial aims to compare perioperative respiratory changes in patients undergoing robot-assisted laparoscopic radical prostatectomy (RALRP) and open radical prostatectomy (ORP). The primary outcome is the change in peak expiratory flow (PEF) from the preoperative period to the early postoperative (2nd hour) period. Secondary outcomes include PEF recovery at 24 hours, and correlations between PEF change and intraoperative factors such as Trendelenburg angle, pneumoperitoneum duration, and ventilatory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male, 18-80 years old
* ASA physical status I-III
* Scheduled for open or robot-assisted radical prostatectomy
* Able to provide informed consent and follow Turkish instructions

Exclusion Criteria:

* Moderate/severe COPD (GOLD II-IV)
* Active upper respiratory tract infection
* Severe OSA requiring CPAP
* Inability to perform standardized PEF maneuver
* Emergency surgery
* Cognitive impairment preventing participation

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in PEF (L/min) | From preoperative baseline to postoperative 2nd hour
  Difference between preoperative and early postoperative PEF values.

SECONDARY OUTCOMES:
Change in PEF from preoperative to postoperative 24th hour | From preoperative measurement (baseline) to postoperative 24th hour
  Evaluates recovery of PEF compared to baseline.
Intraoperative parameters correlated with PEF reduction | From induction of anesthesia to end of surgery
  Correlation between PEF change and intraoperative variables including Trendelenburg angle/duration, pneumoperitoneum pressure/duration, ventilatory pressures, and intraoperative fluid balance.
Incidence of respiratory complications | Within the first 24 hours after surgery
  Frequency of postoperative respiratory events such as desaturation, need for reintubation, or presence of chemosis.

CONTACTS AND LOCATIONS:
Overall Officials: betül aytaç, Principal Investigator — Ankara Bilkent City Hospital, Department of Anesthesiology
Locations (1):
- Ankara Bilkent City Hospital, Department of Anesthesiology, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided